CLINICAL TRIAL: NCT05865041
Title: A Parallel Group Treatment, Phase 2a, Double-blind, Two-arm Study to Investigate the Efficacy and Safety of Farudodstat Tablets Compared With Its Placebo in Male or Female Alopecia Areata Participants Aged 18 Years and Older With 30% or Greater Scalp Hair Loss
Brief Title: Investigate the Efficacy and Safety of Farudodstat Compared With Its Placebo in Adult Alopecia Areata Participants
Acronym: FAST-AA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASLAN003-004
Record Dates: First submitted 2023-04-15; First posted 2023-05-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Alopecia Areata
Keywords: farudodstat; alopecia areata; DHODH inhibitor; ASLAN003
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Intervention Model Description: Approximately 60 participants will be randomized in into one of two treatment sequences:
  * Sequence one: Farudodstat 100mg twice daily for 12 weeks followed by placebo twice daily for 12 weeks
  * Sequence two: Placebo twice daily for 12 weeks followed by farudodstat 100mg twice daily for 12 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Farudodstat for 12 weeks followed by placebo for 12 weeks (Experimental): Farudodstat 100mg twice daily for 12 weeks followed by matching Placebo twice daily for 12 weeks
  Interventions: Drug: Farudodstat; Drug: Placebo
- Placebo for 12 weeks followed by farudodstat for 12 weeks (Experimental): Matching Placebo twice daily for 12 weeks followed by farudodstat 100mg twice daily for 12 weeks
  Interventions: Drug: Farudodstat; Drug: Placebo

INTERVENTIONS:
Drug: Farudodstat — Farudodstat tablets administered orally
  Other Names: ASLAN003
Drug: Placebo — Placebo tablets administered orally
  Other Names: Placebo Comparator

SUMMARY:
The main purpose of this study is to measure the efficacy of farudodstat compared to placebo at Week 12 from the treatment start, in adult participants with Alopecia Areata (AA) with 30% or greater scalp hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age and a weight of ≥40 kg at the time of signing the informed consent)
* Moderate, severe, or very severe Alopecia Areata (AA), as determined by meeting the following criteria:

  1. Clinical diagnosis of AA with no other etiology of hair loss (e.g., telogen effluvium, androgenetic alopecia, etc.)
  2. At least 30% scalp hair loss, as defined by a SALT score ≥30
  3. Current episode of hair loss lasting at least 6 months and not exceeding 7 years at the time of Screening. Participants who have AA for longer than 7 years may be enrolled if episodes of regrowth, spontaneous or under treatment, have been observed on the affected areas over the past 7 years
  4. No appreciable change (i.e., change exceeding 20 points on SALT score) in terminal hair regrowth within 6 months

Exclusion Criteria:

* Known history of androgenic alopecia or female pattern hair loss prior to AA
* Other types of alopecia (including, but not limited to traction and scarring alopecia, telogen effluvium, diffuse type of AA)
* History or presence of hair transplants
* Other scalp disease that may impact AA assessment or require topical treatment (including, but not limited to scalp psoriasis, seborrheic dermatitis, actinic keratosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-09-12 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of change from baseline in Severity of Alopecia Tool (SALT) score at Week 12 from the treatment start. | Treatment Start to Week 12
  The Severity of Alopecia Tool (SALT) is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss).
Incidence of adverse events (AEs) up to Week 28 | Treatment Start to Week 28
Number of participants with clinically significant laboratory parameters | Treatment Start to Week 28
Number of participants with clinically significant Electrocardiogram (ECG) parameters | Treatment Start to Week 28

SECONDARY OUTCOMES:
Change from baseline in Severity of Alopecia Tool (SALT) score at Week 12 from the treatment start. | Treatment Start to Week 12
  The Severity of Alopecia Tool (SALT) is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss).
Proportion of participants achieving Severity of Alopecia Tool (SALT) ≤20 at Week 12 from the treatment start. | Treatment Start to Week 12
  The Severity of Alopecia Tool (SALT) is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss).
Proportion of participants achieving 50% Improvement of Severity of Alopecia Tool (SALT) (SALT50) at Week 12 from the treatment start. | Treatment Start to Week 12
  The Severity of Alopecia Tool (SALT) is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss).
Time to Severity of Alopecia Tool (SALT) score improvement of 50% by Week 12 from the treatment start. | Treatment Start to Week 12
  The Severity of Alopecia Tool (SALT) is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss).
Proportion of participants achieving 75% Improvement of Severity of Alopecia Tool (SALT) (SALT75) at Week 12 from the treatment start. | Treatment Start to Week 12
  The Severity of Alopecia Tool (SALT) is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss).
Time to Severity of Alopecia Tool (SALT) score improvement of 75% by Week 12 from the treatment start. | Treatment Start to Week 12
  The Severity of Alopecia Tool (SALT) is a quantitative assessment of scalp hair loss with scores ranging from 0 (no scalp hair loss) to 100 (complete scalp hair loss).
Proportion of participants with Scalp Hair Assessment Patient Reported Outcome (PRO)™ score of 0 or 1 with a ≥2-point improvement at Week 12 from the treatment start among participants with a score of ≥3 at baseline. | Treatment Start to Week 12
  Participants will assess the severity of their scalp hair loss using 5-point Scalp Hair Assessment PRO™️ scale (0-4) with 4 being the most scalp hair loss
Proportion of participants achieving Clinician Reported Outcome (ClinRO) measure for Eyebrow Hair Loss™ 0 or 1 with ≥2-point improvement from baseline (Among Participants with scores ≥2 at Baseline) at Week 12 from the treatment start. | Treatment Start to Week 12
  ClinRO is scored from 0 to 3 with the 3 representing the most eyebrow hair loss.
Proportion of participants achieving Clinician Reported Outcome (ClinRO) measure for Eyelash Hair Loss™ 0 or 1 with ≥2-point improvement from baseline (among participants with scores ≥2 at baseline) at Week 12 from the treatment start. | Treatment Start to Week 12
  ClinRO is scored from 0 to 3 with the 3 representing the most eyelash hair loss.
Proportion of participants achieving Patient Reported Outcome (PRO) Measure for Eyebrows™ 0 or 1 with ≥2-point improvement from baseline (among participants with scores ≥2 at baseline) at Week 12 from the treatment start. | Treatment Start to Week 12
  Patient's self-assessment of the overall severity of eyebrow hair loss is measured by a 4-point scale (0-3) with photoguide with 3 being the most eyebrow hair loss.
Proportion of participants achieving Patient Reported Outcome (PRO) Measure for Eyelashes™ 0 or 1 with ≥2-point improvement from baseline (among participants with scores ≥2 at Baseline) at Week 12 from the treatment start. | Treatment Start to Week 12
  Patient's self-assessment of the overall severity of eyelash hair loss is measured by a 4-point scale (0-3) with photoguide with 3 being the most eyelash hair loss.
Proportion of participants achieving any amount of hair regrowth at Week 12 after treatment start among participants with alopecia totalis/alopecia universalis (AT/AU) | Treatment Start to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — ASLAN Pharmaceuticals
Locations (19):
- United States (19):
  - 1 Site, Birmingham, Alabama
  - 1 Site, Fountain Valley, California
  - 1 Site, Santa Ana, California
  - 1 Site, New Haven, Connecticut
  - 1 Site, Washington D.C., District of Columbia
  - 1 Site, Coral Gables, Florida
  - 1 Site, Indianapolis, Indiana
  - 1 Site, Louisville, Kentucky
  - 1 Site, Brighton, Massachusetts
  - 1 Site, Minneapolis, Minnesota
  - 1 Site, New Brighton, Minnesota
  - 1 Site, Saint Joseph, Missouri
  - 1 Site, Omaha, Nebraska
  - 1 Site, Cleveland, Ohio
  - 1 Site, Columbus, Ohio
  - 1 Site, Nashville, Tennessee
  - 1 Site, Pflugerville, Texas
  - 2 Sites, San Antonio, Texas
  - 1 Site, Webster, Texas

IPD SHARING:
Plan to Share IPD: No